CLINICAL TRIAL: NCT01170715
Title: Psoriasis Inflammation and Systemic Co-Morbidities: Is it Preventable or Reversible?
Brief Title: Psoriasis Inflammation and Systemic Co Morbidities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, James G. Krueger, MD, PhD, Principal Investigator, Rockefeller University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BDA0688
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Psoriasis
Keywords: Psoriasis; Co morbidities; Inflammation
MeSH Terms: conditions — Psoriasis; Inflammation | interventions — Etanercept

STUDY DESIGN:
Intervention Model Description: Participants will be screened and enrolled based on inclusion/exclusion criteria. Those enrolled will have intervention for 52 weeks and assessed for outcome measures along the way.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Enbrel (etanercept): started with self-injection of 50 mg subcutaneous twice weekly for 12 weeks, followed by self-injection of 50 mg subcutaneous weekly for 40 weeks.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — self-administered for 52 weeks
  Other Names: Enbrel

SUMMARY:
Psoriasis is a chronic relapsing prevalent inflammatory disease affecting 2-4% of the world's population. Severe psoriasis is a disabling disease affecting the physical and emotional well being of patients, and its effect on quality of life is similar to that seen with other major medical diseases such as diabetes, rheumatoid arthritis, and cancer. Lately, it is increasingly being recognized that psoriasis is not merely a skin disease but is probably associated with other co-morbidities such as psoriatic arthritis, Crohn's disease, the metabolic syndrome and cardio-vascular diseases (CVD). The metabolic syndrome is a combination of diabetes mellitus type II (or insulin resistance), hypertension, central obesity, and combined hyperlipidemia (elevated LDL; decreased HDL; elevated triglycerides). As the literature linking psoriasis and the metabolic syndrome expands, also reports of an increased rate of CVD mortality in psoriasis patients accumulates. These data emphasize that metabolic dysregulations are the leading risk factors for occlusive vascular events and early death in patients with severe psoriasis. Progress in understanding the pathogenesis of these apparently diverse diseases has discovered that low-grade systemic inflammation might be the common physiological pathway that may provide the biological plausibility of the associations discovered in the epidemiological studies. Since some of these co-morbidities often become clinically apparent years after the onset of psoriasis we assume that controlling systemic inflammation might prevent or reverse some of these co-morbidities.

Presently there is no study in psoriasis that shows that a "systemic" co-morbidity can be prevented or treated by reversing skin inflammation.

DETAILED DESCRIPTION:
Psoriasis is the most prevalent immune-mediated skin disease affecting 2-4% of the world's population. Severe psoriasis is a disabling disease affecting the physical and emotional well being of patients, and its effect on quality of life is similar to that seen with other major medical diseases such as diabetes, rheumatoid arthritis, and cancer. Psoriasis is a prototypical Th-1 and Th-17 inflammatory disease, which demonstrates a complex interplay between innate and adaptive immunity. Although the etiology of psoriasis in still not completely elucidated, on the basis of existing knowledge, it is obvious that psoriasis is a complex trait involving genetic, metabolic and immune mechanisms as well as environmental factors. Moreover, it is increasingly being recognized that psoriasis is not merely a skin disease but is probably associated with other co-morbidities such as psoriatic arthritis, Crohn's disease, the metabolic syndrome and CVD. Some of these co-morbidities often become clinically apparent years after the onset of psoriasis and are frequently found in patients with severe disease. Furthermore, recently, studies based on large cohorts of psoriasis patients showed that severe psoriasis was association with increased mortality and CVD was found to be the most common cause of death. The metabolic syndrome The metabolic syndrome is a combination of diabetes mellitus type II (or insulin resistance), hypertension, central obesity, and combined hyperlipidemia (elevated LDL; decreased HDL; elevated triglycerides). The prevalence of the metabolic syndrome in the USA is estimated to be up to 15% of the population. Obesity, which is a central feature in the metabolic syndrome, has been termed the modern "epidemic" of the western world. The metabolic syndrome components are associated with increased risk for CVD, which is still the leading cause of death in the western world. Interestingly, inflammation was also implicated in the pathophysiology of the metabolic syndrome. Th-1 and Th-17 cells and cytokines as well as other adipocyte-derived-cytokines adipokines and hormones were identified. Excess numbers of psoriatics are obese, interestingly, the average weight of patients in recent phase 3 studies was around 90Kg. Mechanistic links between psoriasis and its co-morbidities Low-grade inflammation possibly mediated by TNF is suspected to be the biological plausibility explaining the associations discovered in the epidemiological studies linking between psoriasis and its co-morbidities and especially the metabolic syndrome. Progress in understanding the immunology of these apparently diverse diseases has discovered common physiological pathways. Clearly many different tissues and organs have a common blood supply and can be exposed to increased levels of inflammatory cytokines, chemokines and other mediators through the systemic circulation. The "obesity of psoriasis" is thought to be a key link to the metabolic syndrome as well as to CVD. In the past, the only known adipose tissue functions were energy storing and free fatty acids production. However, a dramatic increase of research on the role of adipose tissue has led to the current view that adipose tissue is an active endocrine organ with many secretory products including adipokines and other cytokines. Moreover now it is also being recognized as a part of the innate immune system. Adipocytokines play important roles in the pathogenesis of insulin resistance and associated metabolic complications such as dyslipidemia, hypertension, and premature heart disease. TNF is a major mediator of disrupted insulin receptor signaling. Preventing co-morbidities In view of the chronic nature of the inflammation in psoriasis and the lingering process of metabolic syndrome and CVD development, the most important question is whether effective, long-term control of psoriasis could prevent, reverse, or attenuate these co-morbitides.

Why is this trial important? At present, we do not know how "deep" psoriasis goes as an inflammatory disease.

Inflammatory cells (macrophages) are increased in skin lesions of psoriasis, going as deep as the deep dermis/adipose tissue interface. Macrophages are postulated to be cells increased in adipose tissue that, in conditions of obesity, produce excess TNF and thus directly cause disrupted insulin receptor signaling in adipocytes. The extension of inflammation in skin lesions could well continue into the fat, with common inflammatory circuits then driving both skin disease and obesity/metabolic syndrome that is so common in psoriasis patients.

However, for the purposes of this study, we consider that the adipose tissue in skin is a functional compartment that is distinct from the epidermis and dermis and that production of adipokines and other mediators in the fat compartment can drive not only the metabolic derangements, but also influence the systemic risk of cardiovascular disease. We believe that treatment of inflammation in the primary site of this disease, epidermis and dermis of skin lesions could have corresponding effects on inflammation in other "co-morbid" tissues.

Adipose tissue underlying psoriasis plaques is the most accessible tissue to direct analysis for a reduction in co-morbidity pathophysiology. Interestingly, psoriasis lesion show altered expression of leptin receptors in the "skin" component18 but no studies have been done to compare "skin" vs. adipose tissue. We want to use powerful, high density, arrays and functional imaging studies to assess the degree of inflammation and associated metabolic derangement in fat tissue and then determine the extent to which a reduction in inflammatory circuits in the skin affects the core pathology in fat tissue. Associated biomarker and functional assessments of the cardiovascular tree will provide critical information on whether associated cardiovascular dysfunction can be reversed by treating inflammation in the primary site. If this study is successful, it will not only extend information on the pathophysiology of psoriasis and disease-specific co-morbid risks, but it will also provide guidance on whether long-term effective treatment of inflammation could improve long-term tissue outcomes deeper than the skin. Some of the studies we propose are "firsts" for the study of psoriasis and stand to create new research approaches for psoriasis and other diseases that have similar inflammatory and co-morbid risks. Preliminary Studies Studies in rheumatoid arthritis (RA) patients, another chronic inflammatory disease associated with increased risk for CVD, showed that response to methotrexate treatment is associated with reduction in CVD events and mortality. Biologic treatments for psoriasis, e.g. anti TNF-α (etanercept) or anti p-40 (ustekinumab), have also been shown to reduce C reactive protein (CRP) in short-term trials. A key hypothesis to this study is that the classical TNF pathway (TNF,IL-1,IL-6,IL-8 then the NF kappa B immediate genes) contributes directly to the metabolic alterations in psoriatic patients and that this pathway could also drive systemic inflammation. CRP is produced in the liver in response to IL-6. Many other inflammatory mediators associated with increased CVD risk are made at excess levels in psoriasis lesions and may well contribute to the systemic inflammation burden through release into the circulation. We have used gene arrays and RT-PCR to follow systemic modulation of these CVD related inflammatory molecules in previous studies and will extend this analysis to adipose tissue in this study. However, the question whether long-term effective management of psoriasis can alter the pathophysiology of its comorbid conditions has not been investigated yet.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18years
* Psoriasis affecting Body Surface Area (BSA) ≥ 10% after washout
* No systemic anti psoriatic therapy ≤ 30days
* Plaque type Psoriasis

Exclusion Criteria:

* Overt diabetes (> 135 mg/dL fasting blood glucose on two (2) separate occasions
* Hypertension as defined as a systolic BP > 140 &/or a diastolic pressure > 90. -Cannot be on more then one (1) antihypertensive medication.
* Currently have any known malignancy or have a history of malignancy in the 5 past years excluding basal cell carcinoma.
* S/P Cardiovascular event such as Myocardial infarction, any open heart surgery, stroke or other vascular occlusive event.
* Known allergy to etanercept
* HIV positive
* HBV positive
* HbA1C >7
* Current use of hypoglycemic medication
* Current use of any anticoagulants
* Current use of any anti-inflammatory medications (except inhaled steroids)
* Females of childbearing age who are pregnant or breast-feeding or not using a contraceptive.
* NYHA Class III and Class IV heart failure
* Positive PPD
* History, physical, or laboratory findings suggestive of any other medical or psychological condition that would, in the opinion of the Principal Investigator, make the candidate ineligible for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-07-13 (Actual); Primary Completion 2013-09-09 (Actual); Study Completion 2013-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Krueger, MD, PhD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 29 subjects were screened but only 21 out of this meet inclusion/exclusion criteria and were assigned to the study
Period: Overall Study
Arm/Group | Experimental Group
Started | 21
Completed | 14
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Group
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Histology
Description: To analyze specimens using histology and gene expression before, during, and after treatment.
Time Frame: From baseline, every 3 months, up to one year (52 weeks).
Population: Cell count was never performed
Arm/Group | Experimental Group
Number analyzed (Participants) | 0

2. Primary Outcome: Percentage Change in IL17A Gene Expression
Description: To analyze specimens using histology and gene expression before, during, and after treatment. Percentage Change in IL17A gene expression is the mean of change from baseline divided by mean of baseline and then multiplied by 100: 100*(PostTreatment-Baseline)/Baseline. Both PostTreatment and Baseline values are means but the percentage is a number.
Time Frame: From baseline, every 3 months, up to one year (52 weeks). Except at 9 months. Biopsies were taken at baseline, 3 months, 6 months and 12 months.
Population: 1 participant was not included
Measure: Number; unit: percent change
Arm/Group | Experimental Group
Number analyzed (Participants) | 20
percent change
  3 months (IL17A) | -98.57
  6 months (IL17A) | -99.08
  12 months (IL17A) | -99.66

3. Secondary Outcome: Percentage of Change in IL17A.
Description: To analyze immunological biomarkers of inflammation in the blood using electrochemiluminescence of the MSD systems approach hs-CRP, IL-2 Receptor, Plasminogen activator inhibitor complex (PAI), tissue plasminogen activator (TPA), anti pro BNP, E-selectin, inflammatory cytokines and markers, metabolic markers, vascular markers [IL= interleukin; MMP =Matrix metallopeptidase; ICAM=Inter-Cellular Adhesion Molecule; VCAM= vascular cell adhesion molecule; SAA=Serum amyloid A;GLP-1= Glucagon-like peptide-1;CRP C-Reactive protein. The markers list: IFN-γ, IL-2, IL-4, IL-5, IL-10, IL-12p70, IL-13, IFN-γ, IL-2, IL-4, IL-5, IL-10, IL-12p70, IL-13, MMP- 1, MMP-3 and MMP-9, CRP, sICAM-1, sVCAM-1, SAA, adiponectin, GLP-1,insulin, resistin and other future markers not known at this time.
  Percentage Change in IL17A is the mean of change from baseline divided by mean of baseline and then multiplied by 100: 100*(PostTreatment-Baseline)/Baseline
Time Frame: From baseline, every 3 months, up to one year (52 weeks). Biopsies were taken at baseline, 3 months, 6 months, 9 months and 12 months.
Population: 1 participant was not included
Measure: Number; unit: percent change
Arm/Group | Experimental Group
Number analyzed (Participants) | 20
percent change
  3 months (IL17A) | -150
  6 months (IL17A) | -107
  9 months (IL17A) | -179
  12 months (IL17A) | -111

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Experimental Group
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 6/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=21)
cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
alcohol detox (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=21)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 6 (6)
gum infection (Gastrointestinal disorders) | 1 (1)
joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 2 (2)
insomnia (General disorders) | 1 (1)
biopsy wound infection (Infections and infestations) | 1 (1)
fatigue (General disorders) | 2 (2)
urinary tract infection (Infections and infestations) | 1 (1)
rectal abscess (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes